CLINICAL TRIAL: NCT00624403
Title: LMA ProSeal & I-Gel : a Prospective Controlled Trial
Brief Title: Comparison of Two Type of Laryngeal Mask : I-Gel & LMA ProSeal
Acronym: I-Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY - Clinical Research and Innovation Director (General Director delegation), University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2007/22
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2014-01

CONDITIONS: Endotracheal Intubation
Keywords: Anesthesia; Laryngeal mask airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): LMA ProSeal
  Interventions: Device: Laryngeal mask insertion (LMA ProSeal)
- 2 (Experimental): I-Gel
  Interventions: Device: Laryngeal mask insertion (I-Gel)

INTERVENTIONS:
Device: Laryngeal mask insertion (LMA ProSeal) — Laryngeal mask insertion
  Other Names: LMA ProSeal
  Arms: 1
Device: Laryngeal mask insertion (I-Gel) — Laryngeal mask insertion
  Other Names: I-Gel
  Arms: 2

SUMMARY:
The i-gel is a new supra glottic airway device with a non inflatable cuff and an oesophageal vent. The aim of this study is to compare this device to the LMA ProSeal. The study is approved by the institutional ethic committee. 222 patients will be enrolled in each group. The objectives of the study will be to compare insertion success rate, leak pressure, ventilatory parameters and adverse event rate.

DETAILED DESCRIPTION:
Supraglottic airway devices are now widely used for surgery requiring general anesthesia. Airway devices are safe and their morbidity rate is very low. The i-gel (Intersurgical Ltd, Wokingham, Berkshire, UK) is a new single-use non-inflatable supraglottic airway device that has not been evaluated in a comparative study.

The aim of this study is to compare i-gel with the LMA ProSeal in a randomized study. Anesthesia protocol is standardized. The supraglottic devices are compared in term of insertion success rate, leak pressure, ventilatory parameters and adverse events. The aim is to demonstrate an enhancement in term of insertion success rate and a diminution of the adverse events. Statistical analysis will used percentage, confidence interval and chi 2 or Fischer's exact test for qualitative data. Quantitative data will be analyzed in mean, standard deviation. Comparison will be made with a student t test or a wilcoxon test. P < 0,05 is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 30 kg
* Surgery allowing the use of laryngeal mask as airway management
* Written informed consent

Exclusion Criteria:

* Difficult intubation criteria (defined by French Anesthesia-Reanimation Society)
* Pulmonary disease
* Gastroesophageal reflux antecedent
* Coeliosurgery
* Inhalation risk
* Hiatus hernia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Insertion success rate | At firste attempt of insertion

SECONDARY OUTCOMES:
Perioperative morbidity | Perioperative period
Airway sealing pressure | Once, when efficient ventilation is reached
Accessibility for stomach tube insertion | Juste after laryngeal mask insertion
Fibre-optic grade | After insertion

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie CROS, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Uniersity Hospital, Bordeaux, Bordeaux, France

REFERENCES:
- [Background] Cros AM. [New laryngeal mask airway: easy and evolution to an better safety]. Ann Fr Anesth Reanim. 2006 Aug;25(8):804-5. doi: 10.1016/j.annfar.2006.06.009. Epub 2006 Jul 20. No abstract available. French. PMID 16859880
- [Background] Asai T. Editorial II: Who is at increased risk of pulmonary aspiration? Br J Anaesth. 2004 Oct;93(4):497-500. doi: 10.1093/bja/aeh234. No abstract available. PMID 15361474
- [Background] Cook TM, Lee G, Nolan JP. The ProSeal laryngeal mask airway: a review of the literature. Can J Anaesth. 2005 Aug-Sep;52(7):739-60. doi: 10.1007/BF03016565. PMID 16103390
- [Background] Keller C, Brimacombe J, Kleinsasser A, Loeckinger A. Does the ProSeal laryngeal mask airway prevent aspiration of regurgitated fluid? Anesth Analg. 2000 Oct;91(4):1017-20. doi: 10.1097/00000539-200010000-00046. PMID 11004067
- [Background] Brimacombe J, Richardson C, Keller C, Donald S. Mechanical closure of the vocal cords with the laryngeal mask airway ProSeal. Br J Anaesth. 2002 Feb;88(2):296-7. doi: 10.1093/bja/88.2.296. PMID 11878665
- [Background] Levitan RM, Kinkle WC. Initial anatomic investigations of the I-gel airway: a novel supraglottic airway without inflatable cuff. Anaesthesia. 2005 Oct;60(10):1022-6. doi: 10.1111/j.1365-2044.2005.04258.x. PMID 16179048
- [Background] Cook TM, McKinstry C, Hardy R, Twigg S. Randomized crossover comparison of the ProSeal laryngeal mask airway with the Laryngeal Tube during anaesthesia with controlled ventilation. Br J Anaesth. 2003 Nov;91(5):678-83. doi: 10.1093/bja/aeg239. PMID 14570790
- [Background] Cook TM, Nolan JP, Verghese C, Strube PJ, Lees M, Millar JM, Baskett PJ. Randomized crossover comparison of the proseal with the classic laryngeal mask airway in unparalysed anaesthetized patients. Br J Anaesth. 2002 Apr;88(4):527-33. doi: 10.1093/bja/88.4.527. PMID 12066729